CLINICAL TRIAL: NCT00368420
Title: Validation of a Score of Predictive Factors for Complete Resection in Platinum-sensitive Recurrent Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: AGO Study Group (Other)
Collaborators: Arbeitsgemeinschaft Gynaekologische Onkologie Austria (Other); MITO (Unknown)
Other Study IDs: AGO-OVAR OP.2; AGO DESKTOP OVAR II
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2011-02

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; recurrence; surgery
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to validate a score developed by the AGO-OVAR for complete resection of the tumor

DETAILED DESCRIPTION:
The multicentre retrospective study AGO-DESKTOP OVAR 1 investigated in a multicentre-setting the question of prognostic factors for a successful (i.e. complete) debulking for recurrence. That way, a hypothesis for a score with 3 factors could be developed:

* PS ECOG = 0
* tumor-free after primary surgery (if unknown: FIGO I/II)
* Ascites < 500 ml.

The goal of this study is to evaluate in a prospective multicentre setting, to what extent this retrospectively defined AGO-score has predictive validity. The criterion aimed at is therefore the rate of complete tumor resections if the three score characteristics are present in invasive epithelial platinum-sensitive ovarian-, fallopian tube- or primary peritoneal cancer. This study will be the second in a series of three: (1) hypothesis building for a potential predictive score for resectability, (2) prospective confirmation of the AGO-score, and (3) application of the AGO-score as inclusion criteria for eligible patients in whom a formal comparison of the role of secondary debulking of relapsed ovarian cancer could be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrence of invasive epithelial ovarian-, fallopian tube- or primary peritoneal cancer of any initial stage who have relapsed after a tumor-free interval of at least 6 months after completion of first-line therapy. The same interval applies to patients with second relapse who are enrolled after completed platinum-containing re-induction therapy.
* Women aged > 18 years
* Patients who have given their signed and written informed consent to data transmission and -processing

Exclusion Criteria:

* Patients with non-epithelial tumors as well as borderline tumors
* Patients who undergo second-look surgery or completion surgery after end of chemotherapy or during the interval
* Only for the study collective: patients with second malignancies who have been treated by laparotomy, as well as other neoplasias, if the treatment could interfere with the treatment of relapsed ovarian cancer
* Patients with a third recurrence
* Patients with so-called platinum-refractory tumor, i.e. progression during chemotherapy or recurrence within 6 months after end of former platinum-containing therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recurrence of invasive epithelial ovarian-, fallopian tube- or primary peritoneal cancer of any initial stage who have relapsed after a tumor-free interval of at least 6 months after completion of first-line therapy.
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2006-09; Primary Completion 2008-07 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Harter, Dr., Principal Investigator — Dr. Horst Schmidt Klinik Wiesbaden; Annette Hasenburg, PD Dr., Study Chair — Universitäts-Frauenklinik Freiburg; Andreas du Bois, Prof. Dr., Study Director — Dr. Horst Schmidt Klinik Wiesbaden
Locations (12):
- Universitätskliniken LKH Innsbruck, Innsbruck, Austria
- University Hospitals Leuven, Leuven, Belgium
- Germany (8):
  - Klinikum der Johann Wolfgang Goethe Universität, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - St. Vincentius Kliniken gAG, Karlsruhe
  - Klinikum Landshut gGmbH, Landshut
  - Städtisches Krankenhaus Lüneburg, Lüneburg
  - Klinikum Neumarkt, Neumarkt
  - HSK, Dr. Horst Schmidt Klinik, Wiesbaden
  - Klinikum der Stadt Wolfsburg, Wolfsburg
- Italy (2):
  - Catholic University of Sacred Heart, Campobasso
  - European Institute of Oncology, Milan

REFERENCES:
- [Result] Harter P, Sehouli J, Reuss A, Hasenburg A, Scambia G, Cibula D, Mahner S, Vergote I, Reinthaller A, Burges A, Hanker L, Polcher M, Kurzeder C, Canzler U, Petry KU, Obermair A, Petru E, Schmalfeldt B, Lorusso D, du Bois A. Prospective validation study of a predictive score for operability of recurrent ovarian cancer: the Multicenter Intergroup Study DESKTOP II. A project of the AGO Kommission OVAR, AGO Study Group, NOGGO, AGO-Austria, and MITO. Int J Gynecol Cancer. 2011 Feb;21(2):289-95. doi: 10.1097/IGC.0b013e31820aaafd. PMID 21270612